CLINICAL TRIAL: NCT06568315
Title: Co-administration of Calcium and Multiple Micronutrient Supplements for Maternal and Newborn Hemoglobin and Iron Status: A Randomized Non-inferiority Trial in Burkina Faso and Pakistan
Brief Title: Co-administration of Calcium and Multiple Micronutrient Supplements for Maternal and Newborn Hemoglobin and Iron Status
Acronym: CaMMS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Institut Africain de Santé Publique (African Institute of Public Health) (Unknown); Aga Khan University (Other); Bill and Melinda Gates Foundation (Other); Children's Investment Fund Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00030029; INV036663 (Other Grant/Funding Number: Bill and Melinda Gates Foundation); 1911-04269 (Other Grant/Funding Number: Children's Investment Fund Foundation)
Record Dates: First submitted 2024-08-19; First posted 2024-08-23 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Anemia, Iron Deficiency
Keywords: calcium; iron; supplementation; anemia; pregnancy
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Counseling messages and supplement packaging do not enable masking of participants or study staff with direct participant contact. Laboratory staff measuring the trial's outcomes and investigators will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent MMS / Calcium (Experimental): Daily multiple micronutrient supplement (providing 30 mg iron) taken concurrently with daily calcium supplement (500 mg)
  Interventions: Dietary Supplement: Concurrent multiple micronutrient and calcium supplementation
- Separate MMS / Calcium (Active Comparator): Daily multiple micronutrient supplement (providing 30 mg iron) taken separately from daily calcium supplement (500 mg)
  Interventions: Dietary Supplement: Separate multiple micronutrient and calcium supplementation

INTERVENTIONS:
Dietary Supplement: Concurrent multiple micronutrient and calcium supplementation — Participants counseled to take United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP) multiple micronutrient supplement providing 30 mg elemental iron and calcium supplement providing 500 mg elemental calcium as 1250 mg calcium carbonate together every morning from enrollment through the end of pregnancy
  Arms: Concurrent MMS / Calcium
Dietary Supplement: Separate multiple micronutrient and calcium supplementation — Participants counseled to take United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP) multiple micronutrient supplement (MMS) providing 30 mg elemental iron every morning and calcium supplement providing 500 mg elemental calcium as 1250 mg calcium carbonate every evening from enrollment through the end of pregnancy
  Arms: Separate MMS / Calcium

SUMMARY:
The World Health Organization (WHO) currently recommends the pregnant women receive iron-containing supplements and, in settings where calcium intake is low, calcium supplements. Supplements are to be taken at two separate times of the day as calcium may interfere with iron absorption. The goal of this clinical trial is to learn whether taking daily calcium supplements and iron-containing multiple micronutrient supplements together, at the same time, has any negative impact on the hemoglobin or iron status of pregnant women or the woman's infants. Participants will be randomly assigned and counseled to either take the supplements together every morning or to take the multiple micronutrient supplement in the morning and the calcium supplement in the evening. Participants will visit the antenatal clinic monthly and be asked to provide a blood sample in early, mid, and late pregnancy. Researchers will also take blood samples from infants at the time of birth.

DETAILED DESCRIPTION:
Women of reproductive age in low-and-middle-income countries typically consume diets inadequate in many micronutrients. Resulting micronutrient deficiencies are further exacerbated during pregnancy by the increased demands of the developing fetus. Studies show that antenatal micronutrient supplementation can have important benefits for maternal and infant health. While WHO currently recommends daily iron and folic acid supplementation, many countries are transitioning to multiple micronutrient supplementation (MMS) based on evidence of its further benefit in reducing risk of low birth weight, small-for-gestational age births, stillbirths, and preterm delivery. WHO also recommends calcium supplementation for women in settings where calcium intake is low to reduce high blood pressure and prevent preeclampsia and preterm birth.

Women are instructed to take calcium supplements separately from iron-containing supplements to avoid any negative impact of calcium on iron absorption. However, evidence that calcium limits iron absorption is largely from studies of single test meals. Research on the longer-term implications of consuming the two nutrients together for iron status and hemoglobin is limited, particularly in pregnancy. This is an important research question as limiting the number of times per day that a woman needs to take supplements is likely to improve adherence to the regimen. There is also interest in designing a new MMS formulation that includes calcium such that women could take a single tablet daily.

This individually randomized controlled non-inferiority trial will enroll 1,600 women in both Burkina Faso and Pakistan to assess the impact of co-administering calcium (500 mg elemental calcium as calcium carbonate) and multiple micronutrient supplements (including 30 mg elemental iron), compared with the currently recommended practice of taking the supplements at two separate times of the day, on hematological and iron status of pregnant women and the women's infants. The sample size is based on a non-inferiority margin of -3.0 g/L, 90% power, a one-sided α=0.025, a standard deviation of 17 g/L for the primary hemoglobin outcome, and 15% loss to follow-up.

Potentially eligible women will be identified through antenatal care visits in Burkina Faso and household visits in Pakistan. For those who consent to screening, research staff will measure hemoglobin and conduct a fetal ultrasound exam. Inclusion and exclusion criteria are provided below. Research staff will obtain written documentation of informed consent.

At enrollment, women will be randomized, and research staff will collect socio-demographic data, take anthropometric and blood pressure measurements, and collect a venous blood sample. Women will receive counseling based on the randomly assigned intervention and be given a supply of study supplements. Research staff will see women monthly at antenatal visits to collect information on adherence by recall and pill count, side effects, signs/symptoms of anemia, and information on any iron treatment that women may have received between visits. Iron treatment prescribed by providers outside of the trial will also be abstracted from medical records. At the mid-pregnancy (20<24 weeks) and late pregnancy (30<34 weeks) visits, research staff will take hemoglobin (HemoCue), anthropometric and blood pressure measurements and collect venous blood samples. Women with severe anemia (<70 g/L) will be referred for treatment. Within 72 hours of birth, research staff will collect a heel prick blood sample from infants. Blood samples will be processed at antenatal clinics and transferred to central laboratories for measurement of hematological parameters, iron status, and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Burkina Faso: married or unmarried pregnant women aged ≥15 years
* Pakistan: married pregnant women ≥18 years
* Willing to receive all antenatal care at a study clinic
* Willing to stop iron folic acid supplementation to receive the study intervention
* Hb ≥70 g/L
* 6<20 weeks of gestation based on fetal ultrasound

Exclusion Criteria:

* Burkina Faso: <15 years or unmarried pregnant women <18 years without consent from parent / guardian
* Pakistan: pregnant women <18 years.
* Unwilling to receive antenatal care at a study clinic
* Unwilling to stop iron folic acid supplementation to receive the study intervention
* Hemoglobin < 70 g/L
* <6 weeks of gestation or ≥20 weeks of gestation
* Non-viable or extrauterine pregnancy
* Any contraindications to study supplements

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin concentration of pregnant women | 30<34 weeks of gestation
  Hemoglobin measured by hematology analyzer

SECONDARY OUTCOMES:
Ferritin concentration | 30<34 weeks of gestation
  Ferritin (μg/L)
Soluble transferrin receptor (sTfR) concentration | 30<34 weeks of gestation
  sTfR (mg/L)
Hepcidin concentration | 30<34 weeks of gestation
  Hepcidin (ng/mL)
Erythropoietin (EPO) concentration | 30<34 weeks of gestation
  EPO (mIU/mL)
sTfR-Ferritin index | 30<34 weeks of gestation
  sTfR:log10(ferritin)
Hepcidin-EPO ratio | 30<34 weeks of gestation
  Hepcidin:EPO
Red blood cell (RBC) count | 30<34 weeks of gestation
  RBC count
Mean corpuscular volume (MCV) | 30<34 weeks of gestation
  MCV (fL)
Mean corpuscular hemoglobin (MCH) | 30<34 weeks of gestation
  MCH (pg)
Mean corpuscular hemoglobin concentration (MCHC) | 30<34 weeks of gestation
  MCHC (g/dL)
Hemoglobin concentration of infants | within 72 hours of birth
  Hemoglobin (g/L) measured by HemoCue
Ferritin concentration of infants | within 72 hours of birth
  Ferritin (μg/L)

OTHER OUTCOMES:
Proportion of women with anemia | 30<34 weeks of gestation
  Hemoglobin < 110 g/L
Proportion of women with severe anemia (intervention safety) | 20<24 weeks or 30<34 weeks of gestation
  Hemoglobin < 70 g/L
Proportion of women with iron deficiency | 30<34 weeks of gestation
  Ferritin <15 μg/L (adjusted for inflammation)
Proportion of women with iron-deficient erythropoiesis | 30<34 weeks of gestation
  Elevated sTfR concentration
Proportion of women with iron deficiency anemia | 30<34 weeks of gestation
  Concurrent anemia and iron deficiency
Birth weight | within 72 hours of birth
  Infant's birth weight (g)
Proportion of infants born low birth weight | within 72 hours of birth
  Infant weight <2500 g
Gestational age | within 72 hours of birth
  Gestational age at birth (weeks)
Proportion of infants both preterm | within 72 hours of birth
  Gestational age <37 weeks
Weight-for-gestational age Z-score | within 72 hours of birth
  Calculated using INTERGROWTH-21st standard
Proportion of infants born small for gestational age | within 72 hours of birth
  <10th percentile of weight-for-gestational age using INTERGROWTH-21st standard
Proportion of pregnancies ending in miscarriage | <20 weeks of gestation
  Fetal loss <20 gestational weeks
Proportion of pregnancies ending in stillbirth | ≥20 weeks of gestation
  Fetal loss ≥20 gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Palmer, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- Institut Africain de Santé Publique (African Institute of Public Health), Ouagadougou, Burkina Faso
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available on request by contacting the investigative team.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available after publication of the trial's outcomes
Access Criteria: To be agreed upon with investigators